CLINICAL TRIAL: NCT00240929
Title: A Phase II Randomized, Double-Blind, Two-Period Cross-Over Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Liquid Formulation of Palizvizumab (MEDI-493, Synagis), A Humanized Respiratory Syncytial Virus Monoclonal Antibody, in Children With a History of Prematurity
Brief Title: A Phase II Randomized, Double-Blind, Two-Period Cross-Over Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Liquid Formulation of Palizvizumab (MEDI-493, Synagis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP097
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: -Unhealthy Children With a History of Prematurity
MeSH Terms: interventions — Palivizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MEDI-493 — Active Comparator
  Other Names: Synagis

SUMMARY:
A total of 150 children who meet the entry criteria will be randomized 1:1 to receive one of the following treatment sequence A or B.

DETAILED DESCRIPTION:
Phase II, Double-blind, two-period, cross-over study to be conducted at 20 sites the U.S. A total of 150 children who meet the entry criteria will be randomized 1:1 to receive one of the following treatment sequence: Sequence A (single dose of the liquid formulation on Study Day 0 and a single dose of the lyophilized formulation on Study Day 30) or Sequence B (single dose of the lyophized forumation on Study Day 0 and single dose of the liquid formulation on Study Day 30). Children will be followed for adverse events through 30 days after each injection of study drug and will have blood collected for determination of palivizumab concentrations in serum.

ELIGIBILITY:
Inclusion Criteria:

* The child must have been born at greater than or equal to 35 weeks gestation and be greater than or equal to 6 months of age at the time of randomization (child must be randomized on or before their 6-month birthday)
* The child's parent or legal guardian must provide written informed consent; and
* The child must be able to complete the follow-up visits on Study Days 30 and 60 within the protocol specified windows (±2 days)
* Parent/legal guardian of patient has available telephone access.

Exclusion Criteria:

* Be hospitalized;
* Birth hospitalization > 6 weeks duration;
* Be receiving mechanical ventilation at the time of study entry (including CPAP);
* Bronchopulmonary dysplasia (BPD), defined as history of prematurity and associated chronic lung disease with oxygen requirement for >28 days;
* Congenital heart disease (CHD). (Children with medically or surgically corrected [closed] patent ductus arteriosus and no other CHD may be enrolled.)
* Known renal impairment, hepatic dysfunction, chronic seizure disorder, or immunodeficiency;
* Any of the following laboratory findings in blood obtained within 7 days prior to study entry:
* BUN or creatinine >1.5´ the upper limit of normal for age
* AST (SGOT) or ALT (SGPT) >1.5´ the upper limit of normal for age
* hemoglobin <9.0 gm/dL
* white blood cell count <4,000 cells/mm3
* platelet count <110,000 cells/mm3
* Acute illness or progressive clinical disorder;
* History of recent difficult venous access;
* Active infection, including acute RSV infection;
* Previous reaction to IGIV, blood products, or other foreign proteins;
* Received within the past 120 days or currently receiving IGIV, other immunoglobulin products, or any investigational agents;
* Have ever received palivizumab;
* Currently participating in any investigational study; or
* Previously participated in any investigational study of RSV vaccines or monoclonal antibodies.

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2002-09; Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
adverse events through 30 days after each injection of study drug and will have blood collected for determination of palivizumab concentrations in serum. | Day 30

SECONDARY OUTCOMES:
Adverse events and serious adverse events for 30 days after each injection of study drug. | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Losonsky, M.D., Study Director — "Unaffliliated"
Locations (1):
- Packard Children's Hospital at Stanford, Palo Alto, California, United States